CLINICAL TRIAL: NCT06103071
Title: Effectiveness of Membrane Sweeping on Successful Initiation of Labor and Subsequent Vaginal Birth in Patients With Previous One Cesarean Section.
Brief Title: Role of Membrane Sweeping on Initiation of Labor and Vaginal Birth in Previous Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nida Khan, Principal investigator, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HITEC-IMS
Record Dates: First submitted 2023-09-10; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-01

CONDITIONS: Vaginal Birth After Cesarean Section

STUDY DESIGN:
Intervention Model Description: randomization intervention RCT
Who Masked: Participant
Masking Description: lottery method for selection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sweeping group (Active Comparator): Sweeping group include patients in which membrane sweeping started from 37 weeks and performed weekly till 40 weeks. Intervention is the sweeping of membranes from 37 weeks of gestational amenorrhea.
  Interventions: Procedure: Sweeping of membranes
- Non sweeping group (No Intervention): Non sweeping group include patients in which no sweeping of membranes done. No intervention done.

INTERVENTIONS:
Procedure: Sweeping of membranes — After informed consent all the patients in interventional group will have sweeping of membranes from 37 weeks of pregnancy . It will be repeated weekly till 40 weeks.
  Arms: Sweeping group

SUMMARY:
In Pakistan rate of child birth through cesarean section increased from 3.2% in 1992 to 22% in 2018 .Due to increasing rates of cesarean sections and associated morbidity the investigators should focus to reduce rate of primary cesarean section as well as repeat cesarean with cephalic presentation and singleton pregnancy after previous 1 cesarean section. Therefore, all ladies who underwent previous 1 cesarean section for non-recurrent cause should be considered for vaginal birth. Though studies show that membrane sweeping does promote the onset of labor and avoid need for formal induction of labor for prolonged pregnancy but the effects of membrane sweeping in women with a prior cesarean delivery are largely unknown. This is a randomized controlled trial. Objective of the study was to determine the effect of membrane sweeping on the onset of labor, success of vaginal delivery and neonatal outcome in patients with previous one cesarean section.

DETAILED DESCRIPTION:
World Health Organization suggests that ideally cesarean section rate should not be more than 10% to 15%. The investigators should focus to reduce rate of primary cesarean section as well as repeat cesarean with cephalic presentation and singleton pregnancy after previous 1 cesarean section. Therefore, all ladies who underwent previous 1 cesarean section for non-recurrent cause should be considered for vaginal birth. Though studies show that membrane sweeping does promote the onset of labor and avoid need for formal induction of labor for prolonged pregnancy but the effects of membrane sweeping in women with a prior cesarean delivery are largely unknown. It is reported in literature that there is no significant increase risk to maternal or neonatal outcome with membrane sweeping. The rationale of the study was to compare the effect of membrane sweeping with no sweeping in the successful onset of labor in patients with one previous Cesarean Section so that the investigators can reduce the cesarean section rate. Objective of the study was to determine the effect of membrane sweeping on the onset of labor, success of vaginal delivery and neonatal outcome in patients with previous one cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women willing for vaginal birth after lower segment cesarean section from 37 weeks of gestation to 40 weeks.

  2. Previous one caesarean section for non-recurrent cause 3. Singleton pregnancy 4. Cephalic presentation

Exclusion Criteria:

1. Previous uterine rupture
2. Major degree placenta previa
3. Any medical disorder like PIH, diabetes
4. Bad obstetrics history

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who will have onset of labour till 40 weeks | 4 weeks
  Primary outcome include number of participants who will have onset of labour till 40 weeks between two groups ( sweeping and non sweeping groups )

SECONDARY OUTCOMES:
Number of participants having successful vaginal delivery and number of participants having babies admitted in NICU | 5 days
  It includes how many number of participants will have successful vaginal birth after previous 1 cesarean section and fetal outcome, that is admission in NICU.

CONTACTS AND LOCATIONS:
Overall Officials: Nida Khan, MBBS, FCPS, Principal Investigator — HITEC-Institute of Medical Sciences
Locations (1):
- HIT hospital, Rawalpindi, Punjab Province, Pakistan